CLINICAL TRIAL: NCT02099487
Title: Hypofractionated Imrt (Vmat-Ra) With Temozolomide For Elderly Patients, Unsuitable For Surgery With Newly Diagnosed High Grade Glioma
Brief Title: Hypofractionated Imrt (Vmat-Ra) For Elderly Patients With Newly Diagnosed High Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, M.D., Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1139
Record Dates: First submitted 2014-01-24; First posted 2014-03-31 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2014-01

CONDITIONS: Glioma
Keywords: HGG
MeSH Terms: conditions — Glioma | interventions — Radiation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation (Experimental): To evaluate safety and feasibility of hypofractionated Intensity Modulated Radiotherapy
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — hypofractionated IMRT

SUMMARY:
To assess the effect of IMRT using VMAT rapidarc approach, followed by adjuvant temozolomide on survival and quality of life in elderly, poor performance status patients with newly diagnosed HGG.

DETAILED DESCRIPTION:
Investigators designed this study with the aim to assess the effect of IMRT using VMAT rapidarc approach, followed by adjuvant temozolomide on survival and quality of life in elderly, poor performance status patients with newly diagnosed HGG. The potential advantage of this approach is deliver a more selective irradiation to tumor's target with reducing the dose to normal brain and to allow the delivery of a higher dose, optimizing the therapeutic window.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 70 years
* Karnosky performance status (KPS) ≤60
* Histologically confirmed HGG after tumor biopsy

  * GBM
  * Anaplastic Astrocytoma
  * Anaplastic Oligoastrocytoma
  * Anaplastic Oligodendroglioma without IDH1 mutation and no codeletion 1p19q
* Estimated survival ≥ 3 months.
* Normal liver, Kidney and bone marrow function
* Written informed consent

Exclusion criteria:

* Prior radiation therapy
* Other primary cancer

Exclusion Criteria:

-

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
PFS | one year
  Progression free survival

SECONDARY OUTCOMES:
OS | one year
  Overall Survival

OTHER OUTCOMES:
Toxicity | one year
  Incidence of hematologic and non hematologic severe toxicities (grade III/ IV) will evaluate using NCI-CTCA scale. Late toxicity will evaluate using CTCA 4.2
QoL | one year
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Piera Navarria, MD, Study Director — Humanitas Cancer Center
Locations (1):
- ICH Humanitas Cancer Center, Milan, Lombardy, Italy